CLINICAL TRIAL: NCT03442309
Title: Silver Diamine Fluoride Versus Therapeutic Sealants for the Arrest and Prevention of Dental Caries in Low-income Minority Children
Brief Title: Comparative Effectiveness of School-based Caries Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU College of Dentistry (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Boston University (Other); New York City Department of Health and Mental Hygiene (Other Government)
Responsible Party: Principal Investigator, Richard Niederman, Professor, NYU College of Dentistry
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: i17-00578
Record Dates: First submitted 2018-02-09; First posted 2018-02-22 (Actual); Results first posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Dental Caries; Quality of Life
Keywords: dental caries; caries arrest; caries prevention; quality of life; silver diamine fluoride; sealants; interim therapeutic restorations; student achievement; school attendance
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Intervention Model Description: Two-arm, parallel, non-inferiority cluster randomized trial
Who Masked: Outcomes Assessor
Masking Description: The investigators responsible for analyzing the data for primary outcomes will be masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Simple Prevention (Experimental): One drop (0.05 ml) of silver diamine fluoride (Advantage ArrestTM) solution at 38% concentration (2.24 F-ion mg/dose) will be dispensed per child. Posterior tooth surfaces to be treated will be dried, after which the SDF will be applied with a micro-brush to all asymptomatic carious lesions and to all pits and fissures on bicuspids and molar teeth for thirty seconds. Fluoride varnishes (5% NaF) will then be applied to all teeth.
  Dosage frequency will be twice-yearly.
  Interventions: Device: Silver Diamine Fluoride; Device: Fluoride Varnishes
- Complex prevention (Active Comparator): Pits and fissures on all bicuspids and molar teeth will be sealed with glass ionomer sealants (GC Fuji IX). Glass ionomer sealants (interim therapeutic restorations) will also be placed on all frank asymptomatic carious lesions. Fluoride varnishes (5% NaF) will then be applied to all teeth.
  Dosage frequency will be twice-yearly.
  Interventions: Device: Fluoride Varnishes; Device: Glass Ionomer

INTERVENTIONS:
Device: Silver Diamine Fluoride — Silver diamine fluoride (SDF)
  Other Names: Advantage Arrest
  Arms: Simple Prevention
Device: Fluoride Varnishes — Fluoride varnish (FV)
Device: Glass Ionomer — Glass Ionomer Sealants (GC Fuji IX)
  Arms: Complex prevention

SUMMARY:
Dental caries (tooth decay) is the most prevalent childhood disease in the world. Multiple interventions are available to treat and prevent caries. The aim of the proposed study is to compare the benefit of silver diamine fluoride (SDF) and fluoride varnish versus fluoride varnish and glass ionomer sealants. This study is a five-year, cluster randomized, pragmatic controlled trial conducted in public elementary schools in New York City.

DETAILED DESCRIPTION:
Dental caries is the most prevalent childhood disease in the world and can lead to infection, pain, reduced quality of life, and negative educational outcomes. Multiple prevention agents are available to arrest and prevent dental caries, however little is known of the comparative effectiveness of combined treatments in pragmatic settings. The aim of the presented study is to compare the benefit of silver diamine fluoride and fluoride varnish versus fluoride varnish and glass ionomer therapeutic sealants in the arrest and prevention of dental caries.

This is a longitudinal, pragmatic, cluster randomized, single-blind, non-inferiority trial to be conducted in low-income minority children enrolled in public elementary schools in New York City, New York, United States, from 2018-2023. The primary objective is to assess the non-inferiority of alternative agents in the arrest and prevention of dental caries. Secondary objectives are to assess oral health-related quality of life and educational outcomes. Caries arrest will be evaluated after two years, and caries prevention and secondary outcomes will be assessed at the completion of the study. Data analysis will follow intent to treat, and statistical analyses will be conducted using a two-sided significance level of 0.05.

Notably, the standard of care for dental caries is office-based surgery, which presents multiple barriers to care including cost, fear, and geographic isolation. The simplicity and affordability of silver diamine fluoride may be a viable alternative for the arrest and prevention of dental caries in high-risk children.

ELIGIBILITY:
Inclusion Criteria:

* Any primary school in New York City with a Hispanic/Latino student population greater than 50% and,
* A low-income population (defined as a student receiving free or reduced price lunch) of at least 80%.
* Within participating schools, all children are eligible to participate in the study.

Exclusion Criteria:

* Schools that already have a pre-existing school-based dental health program.
* Within participating schools, exclusion criteria for children include those without informed consent or those with consent but without assent.

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 7418 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Niederman, DMD, Principal Investigator — NYU Langone Health; Ryan R Ruff, PhD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University College of Dentistry, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data could be shared with proper approval from participating organizations for relevant and appropriate requests.

REFERENCES:
- [Derived] Ruff RR, Gawande AA, Xu Q, Barry Godin T. Silver Diamine Fluoride vs Atraumatic Restoration for Managing Dental Caries in Schools: A Cluster Randomized Clinical Trial. JAMA Netw Open. 2025 Jun 2;8(6):e2513826. doi: 10.1001/jamanetworkopen.2025.13826. PMID 40489112
- [Derived] Ruff RR, Barry Godin TJ, Niederman R. Noninferiority of Silver Diamine Fluoride vs Sealants for Reducing Dental Caries Prevalence and Incidence: A Randomized Clinical Trial. JAMA Pediatr. 2024 Apr 1;178(4):354-361. doi: 10.1001/jamapediatrics.2023.6770. PMID 38436947
- [Derived] Ruff RR, Habib R, Godin TB, Niederman R. School-based caries prevention and the impact on acute and chronic student absenteeism. J Am Dent Assoc. 2023 Aug;154(8):753-759. doi: 10.1016/j.adaj.2023.05.007. PMID 37500236
- [Derived] Ruff RR, Barry-Godin T, Niederman R. Effect of Silver Diamine Fluoride on Caries Arrest and Prevention: The CariedAway School-Based Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e2255458. doi: 10.1001/jamanetworkopen.2022.55458. PMID 36757696
- [Derived] Ruff RR, Niederman R. Silver diamine fluoride versus therapeutic sealants for the arrest and prevention of dental caries in low-income minority children: study protocol for a cluster randomized controlled trial. Trials. 2018 Sep 26;19(1):523. doi: 10.1186/s13063-018-2891-1. PMID 30257696

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Schools
Groups:
- Experimental Condition: One drop (0.05 ml) of silver diamine fluoride (Advantage ArrestTM) solution at 38% concentration (2.24 F-ion mg/dose) will be dispensed per child. Posterior tooth surfaces to be treated will be dried, after which the SDF will be applied with a micro-brush to all asymptomatic carious lesions and to all pits and fissures on bicuspids and molar teeth for thirty seconds. Fluoride varnishes (5% NaF) will then be applied to all teeth.
  Dosage frequency will be twice-yearly.
  Silver Diamine Fluoride: Silver diamine fluoride (SDF)
  Fluoride Varnishes: Fluoride varnish (FV)
- Active Control: Pits and fissures on all bicuspids and molar teeth will be sealed with glass ionomer sealants (GC Fuji IX). Glass ionomer sealants (atraumatic restorations) will also be placed on all frank asymptomatic carious lesions. Fluoride varnishes (5% NaF) will then be applied to all teeth.
  Dosage frequency will be twice-yearly.
  Fluoride Varnishes: Fluoride varnish (FV)
  Glass Ionomer: Glass Ionomer Sealants (GC Fuji IX) and atraumatic restorations
Period: Overall Study
Arm/Group | Experimental Condition | Active Control
Started | 3739; 22 Schools | 3679; 24 Schools
Completed | 2063; 20 Schools | 2037; 22 Schools
Not Completed | 1676; 2 Schools | 1642; 2 Schools
Not completed — Lost to Follow-up | 1676 | 1642

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experimental Condition | Active Control | Total
Number analyzed (Participants) | 3739 | 3679 | 7418
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.5 (1.9) | 7.6 (1.9) | 7.6 (1.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1954 | 2052 | 4006
  Male | 1785 | 1627 | 3412
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 88 | 37 | 125
  Black | 650 | 596 | 1246
  Hispanic | 1766 | 1882 | 3648
  White | 86 | 67 | 153
  Multiple | 67 | 47 | 114
  Other | 56 | 34 | 90
  Unreported | 1026 | 1016 | 2042
Number of participants with untreated tooth decay [Count of Participants; unit: Participants] — Any instance of tooth decay regardless of severity or number of teeth affected
  Participants | 1016 | 964 | 1980

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With All Caries Arrested
Description: For any participants with any untreated dental caries on teeth at baseline treated with SDF/FV or Glass ionomer/FV to arrest (control) the infection, what is the proportion of subjects that stayed arrested. Differences were compared to the pre-established non-inferiority margin (10%). NOTE: this analysis conducted after COVID-19 suspensions, thus patient enrollment for this outcome is a subset of the total enrollment reported in Participant Flow. It reflects the total enrollment prior to COVID-19 suspensions (N=1398).
Time Frame: Two years
Population: The study was suspended after initial enrollment and treatment in response to COVID-19. The number of subjects for this outcome subsequently reflects only those enrolled before COVID-19 suspensions and successfully completed a follow-up procedure two years later.
Measure: Count of Participants; unit: Participants
Arm/Group | Experimental Condition | Active Control
Number analyzed (Participants) | 193 | 220
Participants | 108 | 101
Statistical Analysis 1: Comparison: Experimental Condition vs Active Control; Test type: Non-Inferiority — NI margin for arrest difference of 10%; Mean Difference (Final Values) = -.11, 95% CI 2-sided [-.22 to 0.01]

2. Primary Outcome: Prevalence of Dental Caries as Measured by a Clinical Oral Examination
Description: We assessed the prevalence of dental caries through up to four years of follow-up using generalized mixed effects models, with predictors included for time and treatment. Outcomes were assessed comparing the odds of dental caries in participants receiving the active control to those receiving the experimental condition and compared to the pre-established non-inferiority margin.
Time Frame: Participants were evaluated biannually over a total of four years or until lost to follow-up, whichever occurred first.
Measure: Number; unit: # of caries per 1000 tooth years
Arm/Group | Experimental Condition | Active Control
Number analyzed (Participants) | 2063 | 2037
# of caries per 1000 tooth years | 10.2 | 9.8
Statistical Analysis 1: Comparison: Experimental Condition vs Active Control; Test type: Non-Inferiority — Non-inferiority OR (OR δ, 0.63); Odds Ratio (OR) = 0.94, 90% CI 2-sided [0.82 to 1.08]

3. Secondary Outcome: Oral Health-Related Quality of Life
Description: A subset of participants in each treatment group were randomly selected to complete an oral health-related quality of life (OHRQoL) instrument (name: Child Oral Health Impact Profile - Short Form, COHIP-SF19) to compare quality of life pre/post treatment and between treatment groups. Here the differences in COHIP-SF scales are reported six months after initial treatment. After this, COVID-19 suspensions removed any further follow-up for this outcome, which is also why the same sizes are not the same for the full trial. In this analysis, higher scores indicate worse OHRQoL.
  The COHIP-SF scale consists of 19 items. Each item on the scale was scored between 0-3, for a total scale range of 0 to 57.
Time Frame: Six months after initial treatment.
Population: The study was suspended after initial enrollment and treatment in response to COVID-19. The number of subjects for this outcome subsequently reflects only those enrolled until initial suspension and randomly selected to complete the COHIP-SF scale.
Measure: Mean (Standard Deviation); unit: Total COHIP-SF score
Arm/Group | Experimental Condition | Active Control
Number analyzed (Participants) | 111 | 49
Total COHIP-SF score | 14.62 (11.90) | 16.47 (11.09)

4. Secondary Outcome: School Attendance
Description: Annual school attendance (chronic absenteeism) at the school level as recorded by the New York City Department of Education. In evaluating this outcome, we assessed school-level data on the proportion of students who were absent. Additionally, we obtained data from an additional 15 schools which met inclusion criteria but did not participate in the trial as a non-randomized comparison group. This allowed us to compare schools in the experimental group to those in the active control, as well as to a non-randomized untreated group of schools.
Time Frame: 4 years after initial baseline observation
Population: For this outcome schools were assessed for attendance, individual level data was not collected.
Measure: Number (95% Confidence Interval); unit: Beta coefficient comparing exp to ctl
Units Other Than Participants: Schools
Groups:
- Non-treated Schools: Schools that were eligible for the study but not enrolled or randomized
Arm/Group | Experimental Condition | Active Control | Non-treated Schools
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Schools) | 18 | 19 | 15
Beta coefficient comparing exp to ctl | -.037 [-0.062 to -0.011] | -.037 [-0.062 to -0.011] | 0 [0 to 0]

5. Secondary Outcome: Academic Performance
Description: Children participating in schools assigned to each arm of the trial that received care were to have their academic performance evaluated. This outcome was to use academic performance data collected by the school, not investigators.
Time Frame: 4 years after initial baseline observation
Population: Data were not available to be collected due to COVID-19
Arm/Group | Experimental Condition | Active Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Maximum of 4 years of follow-up observation, post-baseline
Arm/Group | Experimental Condition | Active Control
All-Cause Mortality (participants affected / at risk) | 0/3739 | 0/3679
Serious Adverse Events (participants affected / at risk) | 0/3739 | 0/3679
Other Adverse Events (participants affected / at risk) | 0/3739 | 0/3679

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-07-27): https://cdn.clinicaltrials.gov/large-docs/09/NCT03442309/Prot_SAP_002.pdf
  • Informed Consent Form: Recruitment and Informed Consent (2018-02-15): https://cdn.clinicaltrials.gov/large-docs/09/NCT03442309/ICF_001.pdf